

## INFORMED CONSENT FORM

## 

## If you agree, please initial box:

| 1. I confirm that I have read and und sheet version <b>1.0 date 09.09.202</b> opportunity to consider the informathese answered satisfactorily. | 4 for the above study | v. I have had the | |
|---|---|---|---|
| 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. I am aware that I will not be infor until the study has completed. | med which group of | the study I am in | |
| 4. I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from the Sponsor, from regulatory authorities and from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 5. I agree to my General Practitioner being informed of my participation in the study | | | |
| 6. I agree to take part in this study. | | | |
| Name of Participant | Date | Sigr | nature |
| Name of Researcher | Date | Sigr | nature |

Three copies required: one for the patient, one for the researcher and one for hospital case notes.